CLINICAL TRIAL: NCT00879528
Title: Consolidation PET-based and Donor-based After Salvage Therapy in Patients With Hodgkin Lymphoma in Relapse or Refractory
Brief Title: Consolidation PET-based and Donor-based After Salvage Therapy in Patients With HL in Relapse or Refractory
Status: Terminated | Type: Observational
Why Stopped: Failure of accrual achievement
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: IIL-HD0802
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Hodgkin's Lymphoma
Keywords: Hodgkin's Lymphoma; stem cell reinfusion
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Patients with negative PET after salvage therapy — All patients included in the study will treat with a salvage scheme according to each center.
  After the end of salvage therapy, consolidation depends on the outcome of PET:
  PET negative: These patients will follow a standard treatment that includes high-dose chemotherapy with reinfusion of autologous peripheral stem cells.
Other: Patients with positive PET after salvage therapy — All patients included in the study will treat with a salvage scheme according to each center.
  After the end of salvage therapy, consolidation depends on the outcome of PET
  PET positive, the consolidation therapy consists of 2 phases:
  * phase1:common to all consists in a series of high-dose chemotherapy with Melphalan 200 mg/sqm, followed by reinfusion of autologous peripheral stem cells
  * phase2:depends on the availability of a compatible donor. If there is a donor, the patient will continue with an allogeneic transplant preceded by a reduced intensity conditioning.
  If there is not a donor, the patient will continue with a second round of high-dose chemotherapy with BEAM with reinfusion of autologous peripheral stem cells.

SUMMARY:
PET-based consolidation and donor-based therapy after rescue in patients with Hodgkin's lymphoma refractory at first line therapy, or relapse early or late, undergone a second line chemotherapy.

DETAILED DESCRIPTION:
This is a prospective observational study in which patients with positive PET scan after salvage therapy are candidates to a sequential scheme "auto-allotransplantation" in case of availability of a donor . In the event of unavailability of a donor , the same patients are candidates for a double high-dose chemotherapy with autologous stem cell support.

ELIGIBILITY:
Inclusion Criteria:

* Patients confirmed Hodgkin's lymphoma at refractory at first line therapy, relapse early or late;
* Age > 18 years;
* Life expectancy > 3 months;
* Cardiac, pulmonary, renal and liver functions with normal range;
* Written informed consent.

Exclusion Criteria:

* Any psychological, familiar or geographical conditions that could potentially hinder the compliance to the protocol;
* renal failure as creatinine> 1.2 mg/dl or creatinine clearance <60 ml/min;
* AST/ALT or bilirubin> 2.5 times the norm;
* HCV positivity with signs of ongoing viral replication (HCV PCR + AST>1.5-2x normal);
* Heart disease clinically significant: eg. severe hypertension not controlled, multifocal uncontrolled cardiac arrhythmias, symptomatic ischemic heart disease or congestive heart failure class NYHA class III-IV (Annex 2), previous acute myocardial infarction;
* Ventricular ejection fraction <45%;
* decompensated diabetes mellitus not controlled by insulin therapy; Disease with significant pulmonary function defined as FEV1 <65% of predicted or DLCO <50% of predicted value;
* HIV positive patients;
* Patients with uncontrolled infection;
* Neoplasia in the last 3 years except carcinoma in situ uterus, neck and basal skin cancer or prostate cancer in early stage localized exeresi treated with surgery or brachytherapy with curative intent, a good prognosis DCIS breast treated with surgery alone;
* Drug addiction or alcoholism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients confirmed Hodgkin's lymphoma at refractory at first line therapy or relapse
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Patients with negative PET after salvage therapy. To assess prospectively the overall survival and progression-free | 3 years
Patients with positive PET after salvage therapy. Evaluate the role of allogeneic transplantation in these patients after salvage chemotherapy and compare the results with those obtained by 2 cycles of high dose chemotherapy with stem cell | 3 years

SECONDARY OUTCOMES:
Evaluate the percentage of complete remission. | 3 years
Evaluate the haematological toxicity and non-haematological (including acute and chronic GVHD, infections). | 3 years
Evaluation of the chimera. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Luca Castagna, MD, Study Director — Istituto Clinico Humanitas, Dipartimento di Oncologia e Ematologia; Armando Santoro, MD, Study Director — Istituto Clinico Humanitas, Dipartimento di Oncologia e Ematologia
Locations (39):
- Italy (39):
  - Istituto di Ematologia e Oncologia Medica, Policlinico S. Orsola, Bologna, Bologna
  - Unità funzionale di Ematologia AOU Careggi, Florence, Firenze
  - Dipartimento di Oncologia Medica ed Ematologia Istituto Clinico Humanitas, Rozzano, Milano
  - Ematologia Policlinico San Matteo, Pavia, Pavia
  - Ematologia Ospedale S. Maria delle Croci, Ravenna, RA
  - Div Ematologia A.O. Bianchi - Melacrino - Morelli, Reggio Calabria, RC
  - Ematologia Fondazione del Piemonte per l'Oncologia - IRCCS, Candiolo, Torino
  - S.C. Oncologia Medica III Osp. di Circolo, Busto Arsizio, Varese
  - UO di Oncologia Medica e Oncoematologia ASL 14 VCO di Verbania, Verbania, Verbania
  - SC Ematologia - A.O.SS. Biagio, Antonio e Cesare Arrigo, Alessandria
  - SC Enatologia e Trapianto emopoietico AORN San G.Moscati, Avellino
  - Centro di Riferimento Oncologico - Oncologia Medica A, Aviano (PN)
  - Azienda Ospedaliera Policlinico di Bari, Bari
  - Ematologia Spedali Civili, Brescia
  - Presidio Ospedaliero A.Perrino - Divisione di Ematologia, Brindisi
  - Ematologia Ospedale A.Businco, Cagliari
  - SC Ematologia ASO S. Croce e Carle, Cuneo
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.), Meldola (FC)
  - SC Ematologia Azienda Ospedaliera Papardo Nesima, Messina
  - Ematologia Ospedale Niguarda Cà Granda, Milan
  - Unità Linfomi - Dipartimento Oncoematologia Istituto Scientifico S. Raffaele, Milan
  - Centro Oncologico Modenese, Modena
  - AOU Federico II di Napoli, Napoli
  - SCDU Ematologia AOU Maggiore della Carità, Novara
  - ASL 3 Nuoro, UOC Ematologia e CTMO HSF, Nuoro
  - UO Ematologia Ospedale Civile G.da Saliceto, Piacenza
  - Ospedale degli Infermi - Ematologia, Rimini
  - Istituto Regina Elena IFO, Roma
  - Univeristà La Sapienza, Roma
  - Università Cattolica Policlinico Gemelli - Cattedra di Ematologia, Roma
  - UOC Ematologia Ospedale S.Eugenio, Roma
  - Casa sollievo della Sofferenza, San Giovanni Rotondo
  - UOC Ematologia e Trapianti AO Universitaria senese, Siena
  - SC Oncoematologia Azienda Ospedaliera S. Maria di Terni, Terni
  - SC Ematologia Ospedale San Giovanni Battista - Molinette, Torino
  - ASL BAT 1 Divisione di Ematologia, Trani
  - A.O.Cardinale Panico Ematologia e centro trapianti, Tricase (LE)
  - Clinica Ematologica ASUI Integrata di Udine, Udine
  - Oncologia Medica Ospedale di Circolo e Fondazione Macchi, Varese